CLINICAL TRIAL: NCT02298140
Title: Responding to Efficacy Decay Analysis of Artemisinin Based Combination Therapy (ACTs) in Rural Tanzania: Intervening on Provider Compliance and Patient Adherence to Correct Malaria Treatment
Brief Title: Providers' Compliance to Malaria Treatment
Acronym: (PCMT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ifakara Health Institute (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3245
Record Dates: First submitted 2014-07-01; First posted 2014-11-21 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Malaria
Keywords: SMS reminders; Provider's compliance; malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SMS reminders (Experimental): This arm will receive automated mobile phone text message reminders for health workers in outpatient departments of public and private health facilities on issues related to care of malaria patients and suspected patients.
  Interventions: Other: SMS reminders

INTERVENTIONS:
Other: SMS reminders — Text-message reminders about malaria case management will be prepared and distributed to all health workers seeing outpatients in the selected health facilities through their personal mobile phones and facility phones. These messages will reflect ACT recommendations from Tanzania's national guidelines for the diagnosis and treatment of malaria and training manuals. The intervention will run for three months, two text message a day will be send to all identified health workers during regular working hours (i.e. between 8 am to 3 pm), three times a week. To avoid health worker's fatigue of receiving these messages, the messages will also contain some non-malaria humorous, inspirational, motivational and educative contents.
  Other Names: Post training reinforcement

SUMMARY:
INDEPTH Network Effectiveness and Safety Studies in Africa (INESS) have demonstrated a substantial efficacy decay of Artemisinin based combination therapy (ACT) in Tanzania in 2012 (from efficacy of 98% to effectiveness of 18%). Hence system readiness for control and elimination strategies is severely compromised. Sub-optimal health workers' performance in treating malaria cases was a major contributor to the decay, effecting both treatment and patient adherence. If these quantified system failures remain unchecked it will pose major barrier in achieving malaria control and elimination goals. There is growing evidence that mobile phone text message reminders can improve health workers' compliance and patients' adherence to malaria treatment guidelines. Tanzania has recently harnessed all public sector health worker phones into Short Message System (SMS) platform. The investigators intend to exploit this opportunity in a randomized trial of messages to substantially reduce the decay documented by the INESS platform.

The null hypothesis: Sending automated text message reminders to health workers on malaria diagnosis and treatment recommendations, will not have any effects in the quality of malaria case management.

DETAILED DESCRIPTION:
The baseline assessment of systems effectiveness performed by this team, have done a comprehensive quantitative documentation of efficacy decay for ACTs in real world settings; showing how community and provider's contribute to efficacy decay. The proposed text messages reminder intervention builds up from the recent findings of the Kenyan study which demonstrated an improvement in malaria case management by 24%. This level of improvement in malaria case management, if coupled with other systems interventions to improve timely access to ACT providers, should at least double systems effectiveness. This being the case, health systems in developing countries will be able to address these significant challenges hindering taking the diseases eradication agenda forward. Inappropriate care and untimely access to treatment has been identified as one of important elements for ACTs efficacy decay that in turn continues to pose a serious challenge to achieving malaria eradication.

Goal: The study aim to evaluate using cluster randomized control trial whether mobile phone text messages reminders can improve the quality of malaria case management.

Specific objectives:

1. To develop an automated text messaging system to send reminders to mobile phones of health workers based on Tanzanian malaria treatment guidelines;
2. To evaluate the impact of the intervention on providers' compliance to the National Guidelines for Malaria Diagnosis and Treatment (NGMDT);
3. To evaluate the impact of the intervention on patients adherence to malaria treatment with ACT
4. To evaluate the impact of the intervention on reducing baseline efficacy decay levels.

ELIGIBILITY:
Inclusion Criteria:

Dispensaries and health centers; public and private; operating in Rufiji district that provided outpatient services will be eligible for the study. In the intervention arm facility, all health workers who see and take care of patients at the outpatient department (OPD) will be registered to receive automated SMS as the intervention in this study.

During the evaluation phase, all patients attending the surveyed facilities for initial illness consultation will be eligible for inclusion in the study. Assessment of adherence will be performed to malaria patients (who tested positive) and received ACT for treatment.

Exclusion Criteria:

Due to logistical difficulties, health facilities within the Delta region will be excluded in this study. As well, two hospitals in the district will be excluded in the study since they mostly receive referral patients. Also, hospitals have specialized clinic sections with highly trained staff and their nurses or clinicians may be rotating in different departments, hence there may not be health provider's whose primary duties are on OPD patients alone. In addition, health workers in eligible facilities who do not own a mobile phone will be excluded to receive "SMS" reminders.

During evaluation, all severe cases and hospitalized patients will not be included in the surveys. Assessment of adherence study will exclude non residents of the study area.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 712 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Provider Compliance | 10 months
  Proportion of patients presenting to health provider for initial illness consultation with fever (documented fever or history of fever within 48 hours); who are tested for malaria and prescribed ACT for test positive results or not prescribed any antimalarial for test negative results.

SECONDARY OUTCOMES:
Number of fever patients who received diagnostic test | 10 months
  1) Proportion of fever patients receiving a diagnostic test to rule out/in malaria as per national guidelines.
Number of confirmed malaria patients treated with recommended antimalaria | 10months
  Proportion of malaria patients (fever with a positive test routine and gold standard) treated according to malaria treatment guidelines.
Number of malaria patients who received correct dose of ACT | 10 months
  Proportion of patients who receive a correct dose of ACT based on age and/or body weight for malaria treatment
Number of patients with a negative malaria test who did not receive antimalaria | 10 months
  Proportion of negative tested patients who did not receive antimalarials
Number of afebrile patients who are tested for malaria | 10 months
  Proportion of non-febrile (no fever or no history of fever within 48 hours) patients who are tested for malaria
Number of patients who received counselling messages | 10 months
  Proportion of patients who received recommended counseling messages
Number of patients who completed antimalaria doses as instructed | 10 months
  Proportion of complete and incomplete adherent patients, as prescribed by health worker.

CONTACTS AND LOCATIONS:
Overall Officials: Don de Savigny, PhD, Principal Investigator — Swiss Tropical & Public Health
Locations (1):
- Ifakara Health Institute, Rufiji, Coast Region, Tanzania